CLINICAL TRIAL: NCT02902523
Title: Clinical Trial to Assess the Safety and Pharmacokinetics of HUG116 Tablet and Viread® Tablet in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUG-116 P1
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Healthy
MeSH Terms: interventions — Tenofovir

ARMS (2):
- Viread ® tablet 300mg (Active Comparator): Tenofovir disoproxil fumarate
  Interventions: Drug: Viread® tablet 300mg
- HUG116 tablet 245mg (Experimental): Tenofovir disoproxil
  Interventions: Drug: HUG116 tablet 245mg

INTERVENTIONS:
Drug: Viread® tablet 300mg — Single dose administration(PO) in the fasted state
  Arms: Viread ® tablet 300mg
Drug: HUG116 tablet 245mg — Single dose administration(PO) in the fasted state
  Arms: HUG116 tablet 245mg

SUMMARY:
A randomized, open-label, single-dosing, 2x2 crossover study to compare the safety and pharmacokinetics of HUG116 tablet(Tenofovir Disoproxil) with Viread® tablet(Tenofovir Disoproxil Fumarate) in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Body weight over 55kg, in the range of calculated Ideal Body Weight ± 20%
* Subject without a hereditary problems, chronic disease and morbid symptom
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below.(liver, kidney,digestive system, pulmonary,hematooncology, endocrine, urinary,neurology,mental disorder, skeletomuscular, immunology, otolaryngology,cardiovascular)
* Volunteer who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery(appendectomy, hernioplasty are excluded)
* Volunteer who had hypersensitivity reaction to medicines including Tenofovir
* Volunteer who has genetic disorders such as glucose-galactose malabsorption, Lapp lactose deficiency, galactose intolerance
* Sitting systolic blood pressure > 140mmHg or < 100mmHg, sitting diastolic blood pressure ≥ 90mmHg or < 60mmHg, pulse ≥ 100 beats per minute
* Exceed 2 times the normal range of AST, ALT, Total Bilirubin at screening test
* Have the result of Creatinine clearance is less than 50mL/min(Cockcroft-Gault equation applicable)
* Have the result of serum test(RPR Ab(VDRL), HBsAg, HCV Ab, Anti HIV(AIDS)) is a positive
* History of drug abuse, or a positive urine drug screen
* Having ETC drug or herbal medicines within 2 weeks before first administration or OTC drug or vitamin preparations within a week before first administration
* Participation in any other clinical trial involving investigational drugs within 3 months
* Volunteer who had whole blood donation in 2 months, or component blood donation or transfusion in 1 months
* Regular alcohol consumption(over 21 units/week, 1unit=10g of pure alcohol) or volunteers who cannot abstain from drinking during the study
* Volunteers smoking over 10 cigarettes per day in the last 3 months and taking a surfeit of caffeine(caffeine>400mg per day)
* Subjects with planning of dental treatment (tooth extraction, endodontic treatment etc.) and any surgery (aesthetic operation, laser in-situ keratomileusis, laser assisted sub-epithelial keratomileusis etc.) from signed on an informed consent form to post-study visit
* Any condition that, in the view of the investigator, would interfere with study participation

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC)last of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h
Maximum of concentration(Cmax) of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h

SECONDARY OUTCOMES:
Area Under Curve(AUC)inf of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h
tmax of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h
t1/2β of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h
Clearance/F of Tenofovir | 0h(before administration), 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72h

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Seongnam-si, Gyeonggi-do, South Korea